CLINICAL TRIAL: NCT06241378
Title: FEASIBILITY STUDY OF TELE-REHABILITATION IN WOMEN WITH STRESS URINARY INCONTINENCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnya Ahmed Edrees, physiotherapist omnya edrees, Cairo University
Other Study IDs: TELE-REHABILITATION
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Stress Urinary Incontinence
Keywords: tele-rehabilitation stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with stress urinary incontinence: * A hundred twenty-three female with SUI at least once/ week
  * Patients were recruited from Kasr Al Aieny women's health outpatient clinic, Giza, Egypt.
  * Females with an age range 18-65years.
  * Being able to read and write
  * Being able to use Internet and phone services.
  * All of patients with no history of other neurological manifestation.
  * Primiparous and multiparous women.
  Interventions: Device: perineometer device for physiotherapy

INTERVENTIONS:
Device: perineometer device for physiotherapy — measuring the vaginal pressure for stress urinary incontinence patients

SUMMARY:
Tele-rehabilitation involves health care services, support and information provided remotely via digital communication and devices. It intends to facilitate effective delivery of health services such as physical therapy by improving access to care and information and managing health care resources. Other terms such as telehealth, telemonitoring, tele-rehabilitation, tele-education and tele-assistance describe digital practice. Due to the pandemic caused by coronavirus disease 2019 (COVID-19), health associations worldwide have released recommendations about care from distance using tools of communication and information technologies

DETAILED DESCRIPTION:
The female pelvic floor serves multiple functions: pleasure and sexuality, parturition, urination and urinary continence, defecation and fecal continence, and keeping the pelvic organs in position. To perform its functions, the pelvic floor needs an intact anatomical structure, consisting of muscle, connective tissue, and nerves. Moreover, its function is subject to control by the central nervous system. Pelvic floor function and continence can thus be impaired not only by direct anatomical injury, as in vaginal delivery, but also by dysfunctional neural control, e.g., in neurologic disease, diabetic neuropathy, and cognitive disorders (lange, 2007).

The percentage of women suffering from pelvic floor dysfunction (PFD) ranges from 30% to 50%, the main types of female pelvic floor dysfunction involve urinary and/or fecal incontinence and prolapse of the female reproductive organs. Pregnancy and delivery are an important risk factor for urinary incontinence (jundt et al., 2015).

One of the most problems of pelvic floor dysfunction is stress urinary incontinence (SUI), (SUI) defined as the involuntary, sudden loss of urine secondary to increased intra-abdominal pressure that is bothersome or affecting the patient's quality of life. Physical activities precipitating SUI include laughing, sneezing, straining, coughing, or exercising. Patients may refer to a sudden loss of urine as "leaking," "dripping" or "flooding." The patient may initially present with urinary complaints of frequency, urgency, and dysuria. SUI affects 15.7% of adult women; 77.5% of women report the symptoms to be bothersome and 28.8% report the symptoms to be moderate to severe. Prevalence of SUI increases with age, particularly with menopause (Nygaard et al., 2008).

Stress urinary incontinence can exert a significant impact on a patient's life. Treatment aims at improving the quality of life. Complete resolution of SUI may not be feasible, and a combination of behavioral, pharmacological, and surgical treatment may be necessary. Some patients may be satisfied with improved SUI without complete resolution especially if it avoids surgery.

Tele-rehabilitation involves health care services, support and information provided remotely via digital communication and devices. It intends to facilitate effective delivery of health services such as physical therapy by improving access to care and information and managing health care resources. Other terms such as telehealth, telemonitoring, tele-rehabilitation, tele-education and tele-assistance describe digital practice. Due to the pandemic caused by coronavirus disease 2019 (COVID-19), health associations worldwide have released recommendations about care from distance using tools of communication and information technologies (Dantas et al., 2020).

Although the panadeimic has been decreased, with, tele-rehabilitation. The patient don't have to drive to the doctor's office or clinic, park, walk or sit in a waiting room when he is sick. Everyone can see his doctor from the comfort of his own bed or sofa. Virtual visits can be easier to fit into a busy schedule. With, telerehabilitation. Depending on the patient schedule, NO one will have to take time from work or arrange for child care.

Research question:

This study was done to answer the following question: was it feasible to assess stress urinary incontinence through tele-rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* - Females complaining of stress urinary incontinence for at least once per week.
* An age range of 20-65 years.
* Being able to read and write.
* Primiparous or multiparous women.
* Being able to use the Internet, phone services, and online platforms.

Exclusion Criteria:

Patients will be excluded if they have: - - Pregnancy.

* Previous surgery for treating SUI.
* Malignancy in the lower abdomen/ pelvis.
* Any psychiatric disorder that may affect the cognitive function
* Neurological disease with affected sensation of the legs or lower abdomen
* Neurogenic bladder.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Females complaining of stress urinary incontinence for at least once per week.
  - An age range of 20-65 years.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-27 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the efficacy of tele-rehabilitation in stress urinary incontinence patients | basline
  This study will be carried out to investigate the feasibility of assessing stress urinary incontinence through tele-rehabilitation.

CONTACTS AND LOCATIONS:
Locations (1):
- CU, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abe-Takahashi Y, Kitta T, Ouchi M, Okayauchi M, Chiba H, Higuchi M, Togo M, Shinohara N. Reliability and validity of pelvic floor muscle strength assessment using the MizCure perineometer. BMC Womens Health. 2020 Nov 19;20(1):257. doi: 10.1186/s12905-020-01127-x. PMID 33213429
- [Background] da Mata KRU, Costa RCM, Carbone EDSM, Gimenez MM, Bortolini MAT, Castro RA, Fitz FF. Telehealth in the rehabilitation of female pelvic floor dysfunction: a systematic literature review. Int Urogynecol J. 2021 Feb;32(2):249-259. doi: 10.1007/s00192-020-04588-8. Epub 2020 Nov 11. PMID 33175229
- See also: Related Info — https://doi.org/10.1007/s00192-020-04588-8